CLINICAL TRIAL: NCT02725034
Title: Diagnosis of Gastric Intestinal Metaplasia With High Definition Endoscopy and Optic Enhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2016SDU-QILU-02
Record Dates: First submitted 2016-03-26; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Gastric Intestinal Metaplasia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Active Comparator): Standard endoscopy with a standard biopsy protocol from the five standard biopsy sites following the updated Sydney System including two from the distal antrum (within 2-3cm from the pylorus, greater/lesser curvature), one from the incisura and two from the mid corpus (greater/lesser curvature).
  Interventions: Device: Standard endoscopy
- Group 2 (Experimental): High definition endoscopy with Optic Enhancement targeted biopsies for gastric intestinal metaplasia.
  Interventions: Device: High definition endoscopy with Optic Enhancement

INTERVENTIONS:
Device: Standard endoscopy
  Arms: Group 1
Device: High definition endoscopy with Optic Enhancement
  Arms: Group 2

SUMMARY:
The purpose of this study is to assess whether high definition endoscopy with Optic Enhancement can reduce the biopsy number needed per patient for the detection of gastric intestinal metaplasia without the loss of corresponding diagnostic yield

DETAILED DESCRIPTION:
Gastric intestinal metaplasia is regarded as an important premalignant lesion for intestinal type gastric cancer. Currently, the histological assessment of gastric intestinal metaplasia still relies on the biopsies took from five sites that the updated Sydney System recommended. However, the updated Sydney System biopsy protocol needs more biopsy number and procedure time, for it is unable to satisfy the diagnosis of gastric intestinal metaplasia. Optic Enhancement is a novel image-enhanced endoscopy system. Targeted biopsy protocol based on high definition endoscopy with Optic Enhancement will be possible for the diagnosis of gastric intestinal metaplasia. This study aims to compare the diagnostic yield of gastric intestinal metaplasia from high definition endoscopy with Optic Enhancement targeted biopsies and a standard biopsy protocol and assess whether high definition endoscopy with Optic Enhancement can reduce the biopsy number needed per patient for the detection of gastric intestinal metaplasia without the loss of corresponding diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* patients with dyspeptic symptoms and aged 40 years or older
* or patients with Helicobacter pylori infection, or histologically verified gastric intestinal metaplasia or atrophic gastritis
* or patients with family history of gastric cancer

Exclusion Criteria:

* presence of gastrectomy, acute gastrointestinal bleeding, or known gastric neoplasia
* presence of conditions unsuitable for endoscopy procedure including coagulopathy, impaired cardiopulmonary function , pregnancy or breastfeeding
* inability to provide informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Difference of the detection rate of gastric intestinal metaplasia between high definition endoscopy with Optic Enhancement targeted biopsies and standard endoscopy with standard biopsy protocol in a per-patient analysis | eight months
Difference of the detection rate of gastric intestinal metaplasia between high definition endoscopy with Optic Enhancement targeted biopsies and standard endoscopy with standard biopsy protocol in a per-biopsy analysis | eight months

SECONDARY OUTCOMES:
Number of biopsies needed in per group | eight months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China